CLINICAL TRIAL: NCT00679107
Title: A Prospective, Randomized, Controlled, Multicenter, Pilot Study of the OP-1 Putty in Uninstrumented Posterolateral Fusions
Brief Title: A Prospective Pilot Study of the OP-1 Putty in Uninstrumented Posterolateral Fusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Biotech Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S99-01US
Record Dates: First submitted 2008-05-13; First posted 2008-05-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Degenerative Lumbar Spondylolisthesis
Keywords: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): autogenous bone graft with the addition of OP-1 Putty
  Interventions: Device: Use of OP-1 Putty in Uninstrumented posterolateral fusion
- 2 (Active Comparator): autogenous bone graft alone
  Interventions: Device: Use of OP-1 Putty in Uninstrumented posterolateral fusion

INTERVENTIONS:
Device: Use of OP-1 Putty in Uninstrumented posterolateral fusion — Use of OP-1 Putty in Uninstrumented posterolateral fusion
  Other Names: Uninstrumented posterolateral fusion

SUMMARY:
This study will explore the use of OP-1 Putty in conjunction with surgical treatment for the treatment of spinal decompression and lumbar spinal fusion.

DETAILED DESCRIPTION:
It is postulated that the addition of OP-1 Putty to autogenous bone will prove beneficial in the treatment of patients requiring decompression and lumbar spinal fusion. The Investigational system is intended to stimulate bone growth. It is indicated as an adjunct or a replacement for autograft in spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a diagnosis of Degenerative Lumbar Spondylolisthesis of Grade I or II with Spinal Stenosis demonstrated by medical history, physical examination a n d radiographic imaging.
2. The subject is a candidate for decompression and spinal fusion with the use of autograft from the iliac crest.
3. The subject requires one level lumbar fusion (L-3 to S-1).
4. The subject has a preoperative Oswestry Disability Index of 30-100.

Exclusion Criteria:

1. The subject has active spinal and/or systemic infection.
2. The subject is morbidly obese.
3. The subject has a known sensitivity to any component of the OP-1 Putty.
4. The subject has spinal instability measured on flexion / extension radiographs of greater than 50% translation of the vertebrae and greater than or equal to 20 degrees of angular motion.
5. The subject uses tobacco or nicotine or is prescribed steroids such as cortisone.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1999-06; Primary Completion 2000-12 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Safety, by comparison of the complications and neurological status within the OP-1treatment groups and the control group (autograft alone). | 6 weeks; 3, 6, 9, 12, and 24 months

SECONDARY OUTCOMES:
Efficacy, by comparison of overall fusion success and time to fusion along with pain / function outcome within the OP-1 treatment groups and the control group (autograft alone). | 6 weeks; 3, 6, 9, 12, and 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - New Haven, Connecticut
  - Chicago, Illinois
  - Royal Oak, Michigan
  - Akron, Ohio
  - Philadelphia, Pennsylvania